CLINICAL TRIAL: NCT07294183
Title: The Effect of an Emotion-Focused Intervention Based on Travelbee's Human-to-Human Relationship Model on Emotion Regulation Skills and Well-Being of Individuals With Renal Transplantation
Brief Title: The Effect of Emotion-Focused Intervention on Emotion Regulation and Well-Being of Individuals With Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Esra Çelik, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AkdenizU-HF-EÇ-01
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Renal Transplantation
Keywords: Renal Transplantation; Emotional Regulation; Emotion-Focused Therapy; Psychosocial Care; Psychiatric Nursing
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled experimental study with a pretest, posttest, and follow-up control group research design.
Who Masked: Participant
Masking Description: In this study, a single-blind (individuals with renal transplantation) method will be applied. Individuals will not be told which group they are in during the study, thus ensuring that individuals are blinded to the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): It was planned to implement eight sessions of emotion-focused intervention sessions to the intervention group determined according to the inclusion and exclusion criteria.
  Interventions: Behavioral: Emotion-Focused Intervention
- Control group (No Intervention): No intervention will be made to the control group.

INTERVENTIONS:
Behavioral: Emotion-Focused Intervention — Emotion-Focused Intervention methods will be applied to the intervention group once a week in eight sessions, each lasting an average of 60 minutes. These sessions will begin with the first outpatient follow-up after discharge and will be administered weekly in a designated practice room at the Akdeniz University Hospital Organ Transplant Center.
  Arms: Intervention group

SUMMARY:
The study was designed to evaluate the effects of an emotion-focused intervention based on the Human-to-Human Relationship Model on emotion regulation skills and well-being in individuals who have undergone renal transplantation. This study was designed as a single-blind randomized controlled trial with a pretest, posttest, and follow-up control group design. Based on the data obtained from the study, the impact of an emotion-focused intervention based on the Human-to-Human Relationship Model on emotion regulation skills and well-being in individuals who have undergone renal transplantation will be evaluated.

DETAILED DESCRIPTION:
Chronic diseases are long-term, often lifelong, health problems that seriously impact an individual's quality of life. These diseases require not only medical treatment but also psychosocial support. Chronic diseases such as kidney failure cause physical and psychological challenges.

Renal transplantation is an effective treatment option for individuals with chronic kidney disease. However, the transplant process and its aftermath pose intense emotional challenges for the patient and their family. Patients undergoing transplantation require increased social support mechanisms, which can directly impact the success of treatment. Renal transplantation is considered an emotional experience that can evoke a range of emotions, from relief and gratitude to anxiety and fear. It is believed that using emotion-focused therapy approaches is important for individuals with renal transplantation to recognize their emotions, regulate them, and replace dysfunctional emotions with functional ones. In this context, this study was designed to evaluate the effects of an emotion-focused intervention based on the Human-to-Human Relationship Model on emotion regulation skills and well-being in individuals after renal transplantation. Data from the study, which uses a pretest and posttest control group design, will be collected using the Personal Information Form, the Emotion Regulation Skills Scale, and the Well-Being Scale. Emotion-focused intervention methods will be administered to the intervention group in eight sessions, each lasting approximately 60 minutes per week, while the control group will receive no intervention. The study population will consist of individuals who have undergone organ transplantation at the Akdeniz University Hospital Prof. Dr. Tuncer Karpuzoğlu Organ Transplantation Research and Application Center, and the sample will consist of 56 individuals who have undergone renal transplantation who met the inclusion and exclusion criteria. Data analysis will be done using Social Sciences Statistics Package 29.0. Descriptive statistics will be used to define the sample, using the Student t-test, Mann-Whitney U test, and the Wilcoxon pair test. The study will assess the effectiveness of Emotion-Focused Intervention in this group.

It is anticipated that it will reduce psychosocial symptoms seen in individuals who have undergone renal transplantation and have an impact on their emotion regulation skills and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Having a renal transplant
* Being over 18 years of age
* Being literate

Exclusion Criteria:

* Having any communication disability (reading, hearing, speaking, etc.)
* Participation in another study simultaneously with this study outside of routine clinical practice
* Having another neurological or psychiatric diagnosis affecting cognitive status
* Having previously undergone a renal transplant
* Having undergone multiple organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Skills Scale | six months
  This self-report scale, which aims to measure emotion regulation skills in individuals, consists of a total of 27 items. It has nine subscales: awareness/attention (e.g., "I paid attention to my feelings"), body sensations (e.g., "My physical sensations were a good indicator of how I was feeling"), clarity (e.g., "I was sure of what emotions I was experiencing"), understanding (e.g., "I was aware of why I felt this way"), acceptance (e.g., "I accepted my feelings"), tolerance (e.g., "I felt able to tolerate my negative emotions"), preparedness for confrontation (e.g., "Even though it felt uncomfortable or anxious, I did what I planned"), self-support (e.g., "I supported myself in emotionally stressful situations"), and change (e.g., "I was able to influence my negative emotions"). The score of the scale is calculated based on the total score of the items, and a high score indicates high emotion regulation skills.

SECONDARY OUTCOMES:
Well-Being Scale | six months
  The scale is a self-report measurement tool that assesses participants' perceptions of their well-being and relies on individuals to provide information about themselves. Scale items range from 1 (strongly disagree) to 7 (strongly agree). A total well-being score is obtained by summing the scores of all items. The highest possible score is 56, and the lowest is 8. Higher scores indicate a higher level of well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Esra ÇELİK, Principal Investigator — Akdeniz University Faculty of Nursing
Locations (1):
- Akdeniz University Prof. Dr. Tuncer Karpuzoğlu Organ Transplantation Center, Antalya, Turkey (Türkiye)